CLINICAL TRIAL: NCT01400243
Title: Nicotine for Marijuana Withdrawal
Brief Title: Nicotine Patch for Marijuana Withdrawal
Acronym: NMW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southern Illinois University Carbondale (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NIH/NIDA 1R01DA031006 - 01; R01DA031006 (NIH)
Record Dates: First submitted 2011-03-21; First posted 2011-07-22 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Marijuana Dependence
Keywords: Marijuana; Drug withdrawal symptoms; Nicotine
MeSH Terms: conditions — Marijuana Abuse; Substance Withdrawal Syndrome | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Patch (Placebo Comparator): Placebo patch for 15-day quit period
  Interventions: Drug: Placebo Patch
- Nicotine Patch (Active Comparator): 7 mg Habitrol nicotine patch-15 day quit period
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Nicotine patch 7mg
  Other Names: Habitrol
  Arms: Nicotine Patch
Drug: Placebo Patch — Placebo patch
  Other Names: Placebo patch from Rejuvenations Lab
  Arms: Placebo Patch

SUMMARY:
The purpose of this 3-year trial is to test the efficacy of transdermal nicotine patch versus placebo patch on marijuana withdrawal symptoms in cannabis-dependent individuals, using a randomized, double-blind, and placebo-controlled design. This proposal is in response to RFA-DA-10-016(R01) Medications Development for Cannabis-Related Disorders. Consistent with the goals of this RFA, the overall goal of the proposed project is to assess the impact of transdermal nicotine patch (TNP) on marijuana (MJ) withdrawal (negative affect and craving motivated by negative affect) symptoms in MJ-dependent individuals.

DETAILED DESCRIPTION:
The aim of this proposal is to accurately assess the effects of TNP on MJ withdrawal symptoms across 15 days of biochemically confirmed MJ abstinence using a placebo-controlled, double-blind, randomly assigned treatment design, while closely monitoring any potential adverse effects, including changes in nicotine use and dependence.

To achieve these goals, 116 carefully screened cannabis-dependent individuals (58 female) will be randomly assigned to one of two doses (0 mg or 7mg nicotine) of TNP (transdermal nicotine patch) while they abstain from MJ for 15 days. Subjects will be administered a follow-up phone interview 30 days after the termination of treatment to assess the effects of nicotine-patch treatment on: 1) frequency of nicotine and tobacco smoking intake, 2) Fagerstrom Test of Nicotine Dependence (FTND)-assessed nicotine dependence, 3) new use of nicotine during the time since completion of the study, and 4) marijuana and other drug use patterns. Large financial contingencies will be used to provide a high degree of abstinence and study completion. This will be the first adequately powered study to assess the effects of TNP on MJ negative affect-related withdrawal symptoms and urges to use MJ. Withdrawal patterns and abstinence will be assessed in two groups of MJ-dependent individuals: 1) those who rarely or never smoke tobacco, and 2) those who smoke four or fewer tobacco cigarettes per day (very-light tobacco smokers). A stratified randomization method will be used to control for gender and tobacco-smoker status. It is hypothesized that MJ withdrawal symptoms will be less severe in the group assigned to the 7 mg patch than in the group assigned to the placebo. It is also hypothesized that individuals high in anxiety/neuroticism and those high in aggression/hostility will exhibit greater benefits from TNP than those low in these traits. Given that no gender differences were observed in our preliminary study, gender differences are not predicted. The over-the-counter availability, minimal abuse risks, and minimal adverse side-effects associated with TNP would make it an ideal and highly implementable treatment for MJ dependence if it can be demonstrated to be efficacious in reducing MJ withdrawal symptoms.

ELIGIBILITY:
Inclusion Criteria: Female and male cannabis-dependent MJ smokers aged 18 years or older will be recruited. Inclusion criteria include cannabis dependence as assessed by a Diagnostic and Statistical Manual (DSM-IV)-based structured interview and MJ use on 10-28 occasions per week and be willing to abstain for 15 days. Only individuals who are in good mental and physical health, with a BMI of 17-30 kg/m2, as verified by health questionnaires and the Structured Clinical Interview for DSM-IV (SCID), will participate in this study. Potential subjects will be asked to indicate, on a scale of 1-10, how strong they currently want to quit smoking MJ (from "1" = "not at all" to "10" = "very strong") and will also be assessed with the four-item MJ Stages of Change. Additionally, subjects will fulfill one of two criteria: 1) not smoke or use other tobacco products or 2) smoke tobacco cigarettes or use other nicotine delivery systems (e.g., hookah, cigars, chewing tobacco) fewer than 5 times per day (on average) for the past year. Current use of MJ and tobacco will be verified by detectable urine Tetrahydrocannabinol (THC) and nicotine metabolites. All subjects will be required to provide four pre-quit baseline urine samples. The mean creatinine-normalized THC concentration across these samples must be of 175 ng/ml or greater based. -

Exclusion Criteria:

Criteria include meeting DSM-IV criteria for current abuse or dependence on a substance other than MJ, nicotine, or caffeine, using psychoactive substances (other than MJ, alcohol, nicotine, & caffeine) 6+ times/month, testing positive for stimulants, antidepressants, anxiolytics, and/or opiates (10-panel urine drug test), testing above a salivary cotinine concentration of 150 ng/ml during the initial screening, using creatinine or creatinine-containing supplements, testing positive for adulteration of urine samples, consuming more than 6 alcoholic drinks per day continuously for a month, mental disorders including bipolar disorder, schizophrenia, psychotic symptoms, currently, recently, or ever chronically at significant suicidal risk or experiencing violent thoughts or current major depression. Others that will be excluded include women who are pregnant, lactating, not taking precautions to avoid pregnancy, individuals with significant physical disorders or unstable physical disorders that may represent a severe untreated condition, such as hypertension, as well as those with less than a high school education or equivalent, primary language other than English, and those with significant cognitive impairment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2011-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Gilbert, PhD, Principal Investigator — Southern Illinois University Carbondale
Locations (1):
- Southern Illinois University, Carbondale, Illinois, United States

REFERENCES:
- [Derived] Gilbert DG, Rabinovich NE, McDaniel JT. Nicotine patch for cannabis withdrawal symptom relief: a randomized controlled trial. Psychopharmacology (Berl). 2020 May;237(5):1507-1519. doi: 10.1007/s00213-020-05476-1. Epub 2020 Feb 7. PMID 32034447

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female and male cannabis-dependent individuals 18 years or older were recruited by flyers and advertisements in newspapers to participate in the study in the locally well-know Southern Illinois University Integrative Neuroscience Laboratory and Smoking Lab.
Pre-assignment Details: During four sessions across three weeks prior to quitting the use of marijuana, subjects completed questionnaires that assessed mood, drug use, urge to use marijuana (MJ), questionnaires, and motivation to quit MJ, and provided urine, saliva, and expired breath samples for the level of marijuana and other drug use level.
Period: Overall Study
Arm/Group | Placebo Patch | Nicotine Patch
Started | 64 | 63
Completed | 56 | 52
Not Completed | 8 | 11
Not completed — Protocol Violation | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Patch | Nicotine Patch | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 20.57 (2.43) | 21.19 (3.86) | 20.87 (3.20)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 63 | 127
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 38
  Male | 42 | 47 | 89
Region of Enrollment [Number; unit: participants]
  United States | 64 | 63 | 127

OUTCOME MEASURES:

1. Primary Outcome: Profile of Mood Scale Total Negative Affect (Tension + Depression + Anger)
Description: POMS Total negative affect was assessed during the final pre-quit baseline session and the 8 post-quit sessions (1, 3, 5, 7, 9, 11, 13, and 15 days post-quit). The Total negative affect score has a minimum potential value of "0" = best possibly level and a maximum value of "154" = worst possible level.
Time Frame: 16 days (prequit baseline and 15 days of abstinence)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Patch | Nicotine Patch
Number analyzed (Participants) | 56 | 52
units on a scale
  Baseline POMS Total Negative | 8.52 (1.48) | 8.096 (1.54)
  Post-Quit Day 1 POMS Total Negative | 5.14 (1.66) | 4.615 (1.72)
  Post-Quit Day 3 POMS Total Negative | 6.73 (1.67) | 7.48 (1.73)
  Post-Quit Day 5 POMS Total Negative | 7.86 (1.52) | 6.62 (1.58)
  Post-Quit Day 7 POMS Total Negative | 10.34 (2.45) | 8.60 (2.54)
  Post-Quit Day 9 POMS Total Negative | 7.36 (1.74) | 6.87 (1.8)
  Post-Quit Day 11 POMS Total Negative | 8.30 (1.92) | 7.23 (1.99)
  Post-Quit Day 13 POMS Total Negative | 6.66 (1.64) | 5.31 (1.71)
  Post-Quit Day 15 POMS Total Negative | 6.61 (1.73) | 5.10 (1.80)

2. Secondary Outcome: Patch Guess and Attributions Questionnaire
Description: The Patch Guess and Attributions Questionnaire assesses which type of patch (active versus placebo) the subject believes that he or she was given during the study. This assessment was made at end of treatment (Day 15 of abstinence), the last day on a patch. Scores range from 0 percent to 100 percent chance of being on the nicotine patch for those actually on the placebo patch and from 0 percent to 100 percent chance of being on the nicotine patch for those subjects actually on the nicotine patch. Each subject was asked to indicate the percentage chance that he or she was on the nicotine (as opposed to the placebo) patch. The mean values reported below are the group mean percentage averages.
Time Frame: Day 15 of abstinence
Measure: Mean (Standard Error); unit: Percentage chance on nicotine patch
Arm/Group | Placebo Patch | Nicotine Patch
Number analyzed (Participants) | 56 | 52
Percentage chance on nicotine patch | 49.23 (4.23) | 59.85 (3.59)

3. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: Systolic blood pressure was measured in mmHg during each experimental session prior and subsequent to quitting marijuana.
Time Frame: From baseline to Day 15 of abstinence
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Nicotine Patch | Placebo Patch
Number analyzed (Participants) | 52 | 56
mmHg
  Pre-Quit Baseline SBP | 115.31 (1.72) | 113.48 (1.66)
  Quit-Day 1 SBP | 119.42 (1.82) | 115.21 (1.75)
  Quit-Day 3 SBP | 120.85 (1.74) | 115.00 (1.68)
  Quit-Day 5 SBP | 120.25 (1.82) | 117.64 (1.75)
  Quit-Day 7 SBP | 121.02 (1.91) | 115.77 (1.84)
  Quit-Day 9 SBP | 118.50 (1.75) | 116.73 (1.69)
  Quit-Day 11 SBP | 120.21 (1.85) | 115.80 (1.79)
  Quit-Day 13 SBP | 120.58 (1.68) | 115.63 (1.62)
  Quit-Day 15 SBP | 120.69 (1.78) | 115.07 (1.71)

4. Secondary Outcome: Tobacco and Nicotine Intake
Description: Nicotine intake was assessed by self-reported tobacco cigarettes per month (30 days) at baseline (prior to treatment) and also across the 30 days starting immediately after the end of treatment.
Time Frame: Basesline 30 days prior to study and during the 30 days following the 15-day abstinence phase.
Measure: Mean (Standard Error); unit: Cigarettes per 30 days
Arm/Group | Nicotine Patch | Placebo Patch
Number analyzed (Participants) | 52 | 56
Cigarettes per 30 days
  Pre-Treatment Tobacco/Week | 5.47 (3.28) | 7.75 (3.13)
  Post-Treatment Tobacco/Week | 0.23 (3.87) | 6.66 (3.70)

5. Secondary Outcome: Urinary Tetrahydrocannabinol (THC) Concentration in ng/ml.
Description: Tetrahydrocannabinol (THC) Intake assessed by assessing urine sample creatinine corrected THC in ng/ml urine.
Time Frame: across baseline and at 3, 5, 7, 9, 11, 13, and 15 days of abstinence
Measure: Mean (Standard Error); unit: ng/ml urine creatinine-corrected THC
Arm/Group | Nicotine Patch | Placebo Patch
Number analyzed (Participants) | 52 | 56
ng/ml urine creatinine-corrected THC
  Pre-Quit Baseline THC | 343.35 (78.40) | 400.84 (75.55)
  Post-Quit Day 3 THC | 102.16 (20.43) | 128.49 (19.68)
  Post-Quit Day 5 THC | 61.02 (9.17) | 73.07 (8.83)
  Post-Quit Day 7 THC | 43.86 (6.28) | 54.45 (6.05)
  Post-Quit Day 9 THC | 32.61 (4.35) | 38.25 (4.19)
  Post-Quit Day 11 THC | 26.27 (3.95) | 33.31 (3.81)
  Post-Quit Day 13 THC | 20.04 (2.94) | 27.35 (2.82)
  Post-Quit Day 15 THC | 19.97 (2.88) | 23.70 (2.78)
Statistical Analysis 1: Comparison: Nicotine Patch vs Placebo Patch; Test type: Superiority or Other; p = .05, ANCOVA

6. Secondary Outcome: Heart Rate
Description: Heart rate measured during laboratory assessment sessions.
Time Frame: Baseline through Day 15 of abstinence
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Nicotine Patch | Placebo Patch
Number analyzed (Participants) | 52 | 56
beats per minute
  Pre-Quit Baseline Heart Rate | 65.44 (1.47) | 67.86 (1.42)
  Post-Quit Day 1 Heart Rate | 69.54 (1.46) | 65.98 (1.40)
  Post-Quit Day 3 Heart Rate | 73.0 (1.60) | 68.80 (1.54)
  Post-Quit Day 5 Heart Rate | 73.25 (1.71) | 67.91 (1.65)
  Post-Quit Day 7 Heart Rate | 74.04 (1.65) | 67.34 (1.59)
  Post-Quit Day 9 Heart Rate | 75.83 (1.67) | 69.36 (1.61)
  Post-Quit Day 11 Heart Rate | 73.02 (1.84) | 70.89 (1.78)
  Post-Quit Day 13 Heart Rate | 75.42 (1.64) | 69.88 (1.58)
  Post-Quit Day 15 Heart Rate | 72.50 (1.58) | 70.64 (1.52)
Statistical Analysis 1: Comparison: Nicotine Patch vs Placebo Patch; Test type: Superiority or Other; p < 0.05, ANOVA

7. Secondary Outcome: Diastolic Blood Pressure (DBP)
Description: Diastolic blood pressure measured during each of the experimental sessions-- baseline through 15-days post-quit.
Time Frame: From baseline to Day 15 of abstinence
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Nicotine Patch | Placebo Patch
Number analyzed (Participants) | 52 | 56
mm Hg
  Pre-Quit Baseline DBP | 65.06 (1.27) | 68.05 (1.23)
  Post-Quit Day 1 DBP | 69.94 (1.07) | 68.32 (1.03)
  Post-Quit Day 3 DBP | 72.60 (1.28) | 67.88 (1.24)
  Post-Quit Day 5 DBP | 73.02 (1.21) | 69.46 (1.17)
  Post-Quit Day 7 DBP | 71.62 (1.25) | 68.52 (1.21)
  Post-Quit Day 9 DBP | 70.54 (1.08) | 69.29 (1.04)
  Post-Quit Day 11 DBP | 72.50 (1.17) | 71.57 (1.13)
  Post-Quit Day 13 DBP | 71.19 (1.21) | 70.98 (1.17)
  Post-Quit Day 15 DBP | 72.75 (1.32) | 69.55 (1.27)

8. Primary Outcome: Marijuana Withdrawal Questionnaire (MWC) Total Score
Description: The Marijuana Withdrawal Questionnaire Total Score includes items assessing anxiety, depression, irritability, appetite, aggression/anger, sleep disturbance, somatic disturbances, and craving to use marijuana. The potential range of this total score is from "0" = no withdrawal symptoms to "47" = maximally high levels of withdrawal.
Time Frame: 16 days (prequit baseline and at 1, 3, 5, 7, 9, 11, 13, and 15 days of abstinence)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Patch | Nicotine Patch
Number analyzed (Participants) | 56 | 52
units on a scale
  Pre-Quit Baseline MWC | 4.29 (0.59) | 3.67 (0.61)
  Post-Quit Day 1 MWC | 3.80 (0.53) | 4.35 (0.55)
  Post-Quit Day 3 MWC | 5.16 (0.75) | 7.12 (0.78)
  Post-Quit Day 5 MWC | 5.79 (0.80) | 7.02 (0.83)
  Post-Quit Day 7 MWC | 6.30 (0.84) | 6.98 (0.88)
  Post-Quit Day 9 MWC | 5.64 (0.75) | 6.04 (0.78)
  Post-Quit Day 11 MWC | 5.27 (0.81) | 6.56 (0.84)
  Post-Quit Day 13 MWC | 5.48 (0.76) | 5.23 (0.79)
  Post-Quit Day 15 MWC | 5.11 (0.66) | 5.02 (0.68)

9. Primary Outcome: POMS Vigor/Positive Affect (PA)
Description: Profile of Mood State questionnaire Vigor/Positive Affect scale. The potential range of the Vigor/Positive Affect scale is from "0" (no vigor) to "32" (maximally high vigor score).
Time Frame: 16 days (baseline through day 15 of treatment)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nicotine Patch | Placebo Patch
Number analyzed (Participants) | 52 | 56
units on a scale
  Pre-Quit Baseline Vigor/PA | 12.45 (0.82) | 11.18 (0.79)
  Post-Quit Day 1 Vigor/PA | 12.97 (0.87) | 10.72 (0.84)
  Post-Quit Day 3 Vigor/PA | 13.82 (0.86) | 12.34 (0.83)
  Post-Quit Day 5 Vigor/PA | 14.19 (0.84) | 12.35 (0.81)
  Post-Quit Day 7 Vigor/PA | 14.40 (0.90) | 11.94 (0.86)
  Post-Quit Day 9 Vigor/PA | 14.59 (0.91) | 12.52 (0.88)
  Post-Quit Day 11 Vigor/PA | 14.51 (0.85) | 11.94 (0.82)
  Post-Quit Day 13 Vigor/PA | 14.43 (0.85) | 12.54 (0.82)
  Post-Quit Day 15 Vigor/PA | 15.37 (0.88) | 12.15 (0.85)

ADVERSE EVENTS:
Arm/Group | Nicotine Patch | Placebo Patch
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/64
Other Adverse Events (participants affected / at risk) | 41/63 | 40/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotine Patch (N=63) | Placebo Patch (N=64)
Any nonserious adverse event (General disorders) | 41 | 40
Itchiness at Patch Site (Skin and subcutaneous tissue disorders) | 14 | 6
Redness at patch site (Skin and subcutaneous tissue disorders) | 5 | 5
Nausea (Gastrointestinal disorders) | 10 | 4
Sleep disturbance (Nervous system disorders) | 0 | 5
Headache (General disorders) | 3 | 1
Lucid dreams (General disorders) | 1 | 3
Lightheadedness (General disorders) | 1 | 1
Decreased appetite (General disorders) | 3 | 6
Increased appetite (General disorders) | 0 | 3
Hot or sweating (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The modest sample size limited the ability to precisely characterize how the effects of patch type may be modified by tobacco smoker status, gender, personality traits, and individual differences in marijuana use history.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No